CLINICAL TRIAL: NCT02818582
Title: PREVAIL IV: Double-Blind, Randomized, Two-Phase, Placebo-Controlled, Phase II Trial of GS-5734 to Assess the Antiviral Activity, Longer-Term Clearance of Ebola Virus, and Safety in Male Ebola Survivors With Evidence of Ebola Virus Persistence in Semen
Brief Title: GS-5734 to Assess the Antiviral Activity, Longer-Term Clearance of Ebola Virus, and Safety in Male Ebola Survivors With Evidence of Ebola Virus Persistence in Semen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 999916137; 16-I-N137
Record Dates: First submitted 2016-06-28; First posted 2016-06-29 (Estimated); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2019-10

CONDITIONS: Ebola
Keywords: Liberia; Guinea
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GS-5734 100mg given intravenously daily for 5 days (Active Comparator): Male Ebola survivors with persistent Ebola virus in their semen were given GS-5734 100mg intravenously daily for 5 days
  Interventions: Drug: GS-5734
- Normal saline intravenously for 5 days (Placebo Comparator): Male Ebola survivors with persistent Ebola virus in their semen were given normal saline intravenously daily for 5 days
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: GS-5734 — Daily GS-5734 delivered intravenously (IV) for 5 days
  Arms: GS-5734 100mg given intravenously daily for 5 days
Other: Placebo Comparator — Placebo delivered intravenously (IV) for 5 days.
  Arms: Normal saline intravenously for 5 days

SUMMARY:
Background:

Some people have Ebola virus in their body for months after they recover from Ebola virus disease. Some may have health problems from the virus while others are fine. These people may be able to pass the virus to others. There are currently no drugs for people who have survived Ebola virus disease but still have the virus in their body. A new drug, GS-5734, might help get rid of Ebola virus in semen.

Objective:

To test if GS-5734 helps get rid of Ebola virus in semen and is safe for humans.

Eligibility:

Men who participated in the Ebola survivor study (PREVAIL III) and have evidence of the Ebola virus in their semen

Design:

Participants will be screened with:

Questions

Physical exam

Eye exam

Blood tests

2 semen samples if they have not had it tested recently

Participants must live near the study site in Liberia for 6 months.

Participants will be put into 1 of 2 study groups. They will have an infusion of either GS-5734 or a placebo every day for 5 days. A plastic tube is put into an arm vein. The infusion lasts 1 hour.

Participants will be observed for 1 hour after. They will provide a semen sample on infusion day 4.

After the infusions, participants will have 5 visits in the first month, then 1 per month for 5 more months. These include giving a blood and semen sample.

Blood tests are performed before and after each infusion and the last visit (5 month visit) will also include an eye exam.

When the study is over, if the study drug works and is safe, participants who got the placebo can get the study drug.

DETAILED DESCRIPTION:
With the unprecedented size of the recent 2014-2016 West African Ebola outbreak, the scientific community is learning a great deal about the psychological and physical consequences of Ebola, Ebola viral persistence in survivors, risk of Ebola disease relapse in survivors, and the potential for survivors to transmit the virus to others. Data from PREVAIL III has demonstrated that persistence of Ebola virus in the semen of male survivors is common. In addition to Ebola virus persistence, Ebola relapse causing clinical disease has been well documented.

There are no licensed therapies for the treatment of Ebola virus disease nor for the clearance of persistent Ebola virus in survivors. A safe, effective therapy that can reduce and/or eliminate persistent Ebola virus from semen would reduce the risk of transmission and enable male survivors to resume normal sexual relations without fear of harming loved ones. The mechanism underlying Post-Ebola Syndrome is as yet unknown, but improvement in Post-Ebola signs and symptoms resulting from GS-5734 treatment would be an added benefit.

This study is a double-blind, randomized, two-phase (treatment and longer-term follow-up), two- arm trial of GS-5734 versus placebo among male Ebola survivors with persistent Ebola virus RNA in their semen. Participants are randomized 1:1 to receive either 100 mg of GS-5734 or placebo once daily by intravenous catheter for 5 days. Informed by transaminase elevations in prior Phase I studies in normal healthy subjects, a risk-mitigation strategy includes a built-in dose de-escalation. Participants will be stratified by country and on the basis of one versus two positive semen samples for Ebola virus RNA using the Cepheid GeneXpert platform assessed within 42 days prior to study enrollment. The early Data Safety and Monitoring Board (DSMB) review in August 2016 concluded there was no need for a cohort dose reduction. The protocol expanded to Guinea in October 2017, where the outbreak ended later. Currently there is an outbreak in the Democratic Republic of the Congo where the study team may evaluate conducting this study following the completion of the outbreak.

Antiviral activity, as well as safety and tolerability, will be assessed during the treatment phase. Longer-term clearance of Ebola virus will be assessed during the 5-month follow-up phase. Primary analyses for the assessment of antiviral activity in the treatment phase will focus on the assay negativity rate (ANR; percentage of genital samples that are negative for Ebola) over the first 28 days of the study, as well as clinical and laboratory adverse events. A sample is considered negative by PCR if the test result is undetectable. Primary analysis for the follow-up phase will focus on the ANR collected monthly from months 2 to 6.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals must meet all of the following criteria to be eligible for study participation:

* Men more than or equal to 18 years of age.
* One of two semen samples with Ebola virus RNA detection (defined as a positive PCR for NP or GP using the GeneXpert assay within 42 days prior to randomization).
* Willingness to be available for study evaluations for 6 months.
* Willingness to allow storage of biological samples.
* Willingness to be followed by a Participant Tracker.
* Willingness to refrain from alcohol consumption for study days -7 to 14.
* Willingness to comply with MOH & CDC guidance on using a condom for sexual activity and at least through week 24 of the study.

EXCLUSION CRITERIA:

Individuals meeting any of the following criteria will be excluded from study participation:

* Estimated glomerular filtration rate less than 60 mL/min/1.73m^2
* History of significant renal disease
* History of significant liver disease
* Evidence of liver disease on physical exam such as ascites
* Aspartate transaminase (AST) or alanine transaminase (ALT), greater than the upper limit of normal, a prothrombin time 1.1 times greater than the upper limits of normal, normal, or a total bilirubin > 1.5 times the upper limits of normal(per Division of Acquired Immunodeficiency Syndrome (DAIDS) toxicity tables version 2.0 Nov. 2014).
* Presence of Grade 2 or higher abnormalities for: low hemoglobin, low white blood count (WBC), low platelets, or low or high potassium (per DAIDS toxicity tables version 2.0 Nov. 2014).
* Presence of greater than Grade 2 abnormalities for low or high sodium (per DAIDS toxicity tables version 2.0 Nov. 2014).
* Any condition that, in the opinion of the investigator, would compromise the safety of the study subject or staff, or would prevent proper conduct of the study.

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth S Higgs, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- Partnership of Clinical Research in Guinea (PREGUI) / Centre National de Formation et de Recherche en Santé Rurale de Mafèrinyah, Forécariah, Maferinyah, Guinea
- JFK Hospital Partnership for Research for Vaccines and Infectious Diseases in Liberia (PREVAIL), Monrovia, Liberia

REFERENCES:
- [Background] de Vries DH, Rwemisisi JT, Musinguzi LK, Benoni TE, Muhangi D, de Groot M, Kaawa-Mafigiri D, Pool R. The first mile: community experience of outbreak control during an Ebola outbreak in Luwero District, Uganda. BMC Public Health. 2016 Feb 16;16:161. doi: 10.1186/s12889-016-2852-0. PMID 26883621
- [Background] Bwaka MA, Bonnet MJ, Calain P, Colebunders R, De Roo A, Guimard Y, Katwiki KR, Kibadi K, Kipasa MA, Kuvula KJ, Mapanda BB, Massamba M, Mupapa KD, Muyembe-Tamfum JJ, Ndaberey E, Peters CJ, Rollin PE, Van den Enden E, Van den Enden E. Ebola hemorrhagic fever in Kikwit, Democratic Republic of the Congo: clinical observations in 103 patients. J Infect Dis. 1999 Feb;179 Suppl 1:S1-7. doi: 10.1086/514308. PMID 9988155
- [Background] Feldmann H, Geisbert TW. Ebola haemorrhagic fever. Lancet. 2011 Mar 5;377(9768):849-62. doi: 10.1016/S0140-6736(10)60667-8. PMID 21084112
- [Derived] Higgs ES, Gayedyu-Dennis D, Fischer Ii WA, Nason M, Reilly C, Beavogui AH, Aboulhab J, Nordwall J, Lobbo P, Wachekwa I, Cao H, Cihlar T, Hensley L, Lane HC. PREVAIL IV: A Randomized, Double-Blind, 2-Phase, Phase 2 Trial of Remdesivir vs Placebo for Reduction of Ebola Virus RNA in the Semen of Male Survivors. Clin Infect Dis. 2021 Nov 16;73(10):1849-1856. doi: 10.1093/cid/ciab215. PMID 33709142

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Saline Given Intravenously Daily for 5 Days: Male Ebola survivors with persistent Ebola virus in their semen were given normal saline intravenously daily for 5 days
Period: Overall Study
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Started | 20 | 18
Completed | 20 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days | Total
Number analyzed (Participants) | 20 | 18 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 20 | 18 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 20 | 18 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Assay Negativity Rate (ANR) for Ebola Virus During the Treatment Phase
Description: Mean assay negativity rate (ANR) of semen samples collected during the treatment phase on days 4, 8, 11, 16, 20, 24, & 28. Average of all time points for negative values were compiled for the collected assay values.
  Negativity rate per participant was calculated using all time points by calculating the number of negative results over total number of time points (7). The assay negativity rate was averaged over all participants to get the mean assay negativity rate.
Time Frame: Treatment Phase (assessed at days 4, 8, 11, 16, 20, 24, & 28)
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: proportion of semen samples
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
proportion of semen samples | 0.85 (0.24) | 0.76 (0.3)

2. Primary Outcome: Mean Assay Negativity Rate (ANR) for Ebola Virus During the Follow-up Phase
Description: Mean assay negativity rate (ANR) of semen samples collected during the follow-up phase on weeks 8, 12, 16, 20, & 24. Average of all time points for negative values were compiled for the collected assay values.
  Negativity rate per participant was calculated using all time points by calculating the number of negative results over total number of time points (5). The assay negativity rate was averaged over all participants to get the mean assay negativity rate.
Time Frame: Follow-up phase (assessed on weeks 8, 12, 16, 20, & 24)
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: proportion of semen samples
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
proportion of semen samples | 0.96 (0.1) | 0.81 (0.29)

3. Secondary Outcome: Mean Assay Negativity Rate (ANR) for Ebola Virus During the Treatment Phase
Description: as for outcome 1
Time Frame: Treatment Phase (assessed on days 4, 8, 11, 16, 20, 24, & 28)
Population: Participants who had one of two baseline positive semen sample for Ebola virus
Measure: Mean (Standard Deviation); unit: proportion of semen samples
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 16 | 15
proportion of semen samples | 0.86 (0.24) | 0.86 (0.19)

4. Secondary Outcome: Mean Assay Negativity Rate (ANR) for Ebola Virus During the Treatment Phase
Description: as for outcome 1
Time Frame: Treatment Phase (assessed on days 4, 8, 11, 16, 20, 24, & 28)
Population: Participants who had two of two baseline positive semen sample for Ebola virus
Measure: Mean (Standard Deviation); unit: proportion of semen samples
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 4 | 3
proportion of semen samples | 0.79 (0.25) | 0.28 (0.35)

5. Secondary Outcome: Mean Assay Negativity Rate (ANR) for Ebola Virus During the Follow-up Phase
Description: Mean assay negativity rate (ANR) of semen samples collected during the follow-up phase - weeks 8, 12, 16, 20, & 24. Average of all time points for negative values were compiled for the collected assay values.
  Negativity rate per participant was calculated using all time points by calculating the number of negative results over total number of time points (5). The assay negativity rate was averaged over all participants to get the mean assay negativity rate.
Time Frame: Follow-up phase (assessed on weeks 8, 12, 16, 20, & 24)
Population: Participants who had one of two baseline positive semen sample for Ebola virus
Measure: Mean (Standard Deviation); unit: proportion of semen samples
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 16 | 15
proportion of semen samples | 0.95 (0.12) | 0.9 (0.19)

6. Secondary Outcome: Mean Assay Negativity Rate (ANR) for Ebola Virus During the Follow-up Phase
Description: as for outcome 5
Time Frame: Follow-up phase (assessed on weeks 8, 12, 16, 20, & 24)
Population: Participants who had two of two baseline positive semen sample for Ebola virus
Measure: Mean (Standard Deviation); unit: proportion of semen samples
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 4 | 3
proportion of semen samples | 1 (0) | 0.33 (0.23)

7. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 3.6 (11.94) | -2.22 (7.48)

8. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 2.25 (11.61) | -0.56 (7.25)

9. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 4.05 (12.25) | 10.28 (18.05)

10. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 8.45 (13.2) | 11.78 (20.74)

11. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 13.15 (14.64) | 9.22 (14.97)

12. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 21.45 (21.09) | 4.89 (7.88)

13. Secondary Outcome: Mean Change From Baseline in ALT Value at Day 11
Description: Mean change from baseline in alanine transaminase (ALT) value at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 8.65 (10.91) | 1.78 (8.18)

14. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at day 16
Time Frame: Treatment phase - Day 16
Population: Participants who received intervention and had lab value available at baseline and treatment/follow-up day/week. One subject had missing lab value.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
IU/L | 3.53 (9.06) | -0.06 (8.91)

15. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -0.65 (7.21) | -0.67 (6.89)

16. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 0.4 (10.08) | -2.06 (9.67)

17. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -2.15 (6.28) | -1.22 (7.01)

18. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) Value at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 3.1 (18.29) | -1.78 (8.99)

19. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 5.95 (24.56) | -0.11 (4.56)

20. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -1.55 (8.24) | -1.72 (8.04)

21. Secondary Outcome: Mean Change From Baseline in ALT Value
Description: Mean change from baseline in alanine transaminase (ALT) value at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
IU/L | -0.89 (6.74) | 22.67 (104.56)

22. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 1
Time Frame: Treatment phase - Day 1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | 0.34 (5.13) | 0.24 (2.6)

23. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 2
Time Frame: Treatment phase - Day 2
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | -0.9 (4.28) | -1.45 (2.04)

24. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 3
Time Frame: Treatment phase - Day 3
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | -0.03 (4.28) | -1.42 (3.91)

25. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 4
Time Frame: Treatment phase - Day 4
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | 3.82 (11.84) | -2.24 (2.29)

26. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 5
Time Frame: Treatment phase - Day 5
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | 1.29 (4.63) | -1.24 (4.15)

27. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 8
Time Frame: Treatment phase - Day 8
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | 3.92 (6.43) | 0.34 (2.84)

28. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 11
Time Frame: Treatment phase - Day 11
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | -1.41 (3.6) | -0.17 (2.97)

29. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 16
Time Frame: Treatment phase - Day 16
Population: Participants who received intervention and had lab value available at baseline and treatment/follow-up day/week. Three subjects had missing lab value.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 18 | 17
Seconds | -0.18 (4.76) | 0.26 (4.33)

30. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 24
Time Frame: Treatment phase - Day 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | -0.27 (4.72) | 0.76 (4.2)

31. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention and had lab value available at baseline and treatment/follow-up day/week. Two subjects had missing lab value.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 16
Seconds | 0.52 (3.91) | 0.24 (5.18)

32. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at week 8
Time Frame: Follow-up phase - Week 8
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 17
Seconds | 1.16 (3.65) | 0.62 (3.67)

33. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at week 12
Time Frame: Follow-up phase - Week 12
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | 0.5 (3.95) | 1.29 (3.17)

34. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at week 16
Time Frame: Follow-up phase - Week 16
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 17
Seconds | 0.78 (4.84) | 1.37 (5.22)

35. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at week 20
Time Frame: Follow-up phase - Week 20
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Seconds | 1.83 (5.04) | 0.75 (6.8)

36. Secondary Outcome: Mean Change From Baseline in aPTT Value
Description: Mean change from baseline in activated partial thromboplastin time (aPTT) value at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 31
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 17
Seconds | -0.39 (4.6) | 0.41 (4.7)

37. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) Value at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 2.45 (8.34) | -1.89 (7.38)

38. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) Value at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -0.2 (5.95) | 0.06 (5.56)

39. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 0.35 (6.9) | 10.39 (20.13)

40. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 5.6 (9.08) | 5.72 (15.94)

41. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 8.15 (9.35) | 2.44 (9.51)

42. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 9.4 (12.83) | 1.39 (7.69)

43. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 0.2 (6.87) | -0.22 (8.14)

44. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
IU/L | -1.42 (5.34) | -0.89 (8.38)

45. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -1.25 (5.22) | 0.67 (6.89)

46. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 0.85 (8.6) | -0.83 (9.4)

47. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -1.7 (5.16) | 1.39 (7.91)

48. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate aminotransferase transaminase (AST) value at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 5.85 (24.54) | 1 (8.25)

49. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate aminotransferase transaminase (AST) value at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | 11.4 (36.51) | 1.39 (4.35)

50. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate aminotransferase transaminase (AST) value at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
IU/L | -0.95 (8.91) | -0.67 (8.25)

51. Secondary Outcome: Mean Change From Baseline in AST Value
Description: Mean change from baseline in aspartate transaminase (AST) value at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
IU/L | -1.05 (6.03) | 11.61 (51.06)

52. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.02 (0.15) | 0 (0.13)

53. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.01 (0.08) | -0.01 (0.14)

54. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.03 (0.07) | -0.03 (0.14)

55. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 1.04 (4.16) | -0.06 (0.15)

56. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.13 (0.07) | -0.05 (0.16)

57. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.12 (0.16) | -0.05 (0.15)

58. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.05 (0.18) | -0.03 (0.14)

59. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Ratio | 0.05 (0.19) | -0.05 (0.13)

60. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.06 (0.22) | -0.04 (0.15)

61. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.01 (0.21) | -0.03 (0.19)

62. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | -0.01 (0.24) | -0.18 (0.21)

63. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | 0.04 (0.2) | -0.06 (0.27)

64. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at week 16
Time Frame: Follow-up phase - Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Ratio | 0.09 (0.2) | -0.05 (0.24)

65. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Ratio | -0.05 (0.3) | -0.16 (0.26)

66. Secondary Outcome: Mean Change From Baseline in INR Value
Description: Mean change from baseline in international normalized ratio (INR) value at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Ratio | -0.1 (0.31) | -0.28 (0.2)

67. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.13 (0.51) | 0.22 (0.41)

68. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | 0.09 (0.71) | 0.13 (0.51)

69. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | 0.28 (0.62) | -0.01 (0.62)

70. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | 6.27 (23.42) | -0.24 (0.5)

71. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | 1.28 (0.6) | -0.13 (0.6)

72. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | 0.86 (0.76) | -0.11 (0.65)

73. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.08 (0.56) | 0.04 (0.71)

74. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Seconds | -0.13 (0.84) | -0.17 (0.56)

75. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.1 (0.78) | -0.07 (0.58)

76. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.34 (0.75) | 0.11 (0.61)

77. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.26 (0.59) | -0.27 (0.57)

78. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.22 (0.74) | 0.06 (0.59)

79. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at week 16
Time Frame: Follow-up phase - Week 16
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Seconds | -0.17 (0.59) | -0.03 (0.54)

80. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.25 (0.7) | 0.26 (0.81)

81. Secondary Outcome: Mean Change From Baseline in PT Value
Description: Mean change from baseline in prothrombin time (PT) value at week 24
Time Frame: Follow-up phase - Week 24
Population: Participants who received intervention
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Seconds | -0.41 (0.90) | -0.23 (0.6)

82. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) value at day 1.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (AE) [DAIDS AE grading table] version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

83. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 2.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

84. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 3.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

85. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 4.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 3

86. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 5.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 2 | 2

87. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 5 | 0

88. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 11.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 3 | 0

89. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0

90. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

91. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at day 28.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

92. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at week 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

93. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at week 12.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

94. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at week 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

95. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) Value at week 20.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

96. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for ALT Value
Description: Number of participants with increase in grade from baseline in alanine transaminase (ALT) value at week 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  ALT grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 1

97. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 1.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 1
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 1 | 0

98. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 2.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 2
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 0 | 0

99. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 3.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 3
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 1 | 1

100. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 4.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 4
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 5 | 0

101. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 5.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 5
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 2 | 0

102. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 8
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 2 | 0

103. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 11.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 11
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 0 | 0

104. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 16
Population: as for outcome 29
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 18 | 17
Participants | 1 | 0

105. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 1 | 1

106. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at day 28.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 28
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 16
Participants | 0 | 0

107. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at week 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 8
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 17
Participants | 1 | 1

108. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at week 12.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 12
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 1 | 1

109. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at week 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 16
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 17
Participants | 1 | 2

110. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at week 20.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 20
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 17
Participants | 1 | 2

111. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for aPTT Value
Description: Number of participants with increase in grade from baseline in activated partial thromboplastin time (aPTT) value at week 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  aPTT grade ranges include grade 1 (1.1 - 1.66 x ULN), grade 2 (1.67 - 2.33 x ULN), grade 3 (2.34 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 24
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 17
Participants | 0 | 1

112. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at day 1.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

113. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at day 2.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

114. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) value at day 3.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 4

115. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) value at day 4.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 1

116. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at day 5.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 1

117. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at day 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 3 | 0

118. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) value at day 11.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

119. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at day 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

120. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) value at day 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

121. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at day 28.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

122. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at week 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 1

123. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at week 12.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

124. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at week 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 2 | 0

125. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) value at week 20.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

126. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for AST Value
Description: Number of participants with increase in grade from baseline in aspartate transaminase (AST) Value at week 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  AST grade ranges include grade 1 (1.25-2.5 x ULN), grade 2 (2.6-5.0 x ULN), grade 3 (5.1-10.0 x ULN), & grade 4 (> 10 x ULN)
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 1

127. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 1.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

128. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 2.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

129. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 3.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

130. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 4.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 2 | 0

131. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 5.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

132. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

133. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 11.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

134. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants with increase in grade from baseline in prothrombin time (PT) value at day 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

135. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at day 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

136. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at day 28.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

137. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at week 8.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

138. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at week 12.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

139. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at week 16.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

140. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at week 20.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 1

141. Secondary Outcome: Number of Participants With Increase in Grade From Baseline for PT Value
Description: Number of participants increase in grade from baseline in prothrombin time (PT) value at week 24.
  Lab values were graded using Division of Acquired Immunodeficiency Syndrome (DAIDS) table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE grading table) version 2.0, November 2014 with grade 1 (mild), grade 2 (moderate), grade 3 (severe), and grade 4 (potentially life-threatening).
  PT grade ranges include grade 1 (1.1 - 1.25 x ULN), grade 2 (1.26 - 1.50 x ULN), grade 3 (1.51 - 3.00 x ULN), & grade 4 (> 3.00 x ULN)
Time Frame: Follow-up phase - Week 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

142. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

143. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

144. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 5

145. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 3

146. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 2 | 2

147. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 4 | 0

148. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 3 | 0

149. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0

150. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

151. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

152. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

153. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

154. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

155. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

156. Secondary Outcome: Participants With Grade 1 ALT Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) alanine transaminase (ALT) level at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0

157. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

158. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

159. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 4

160. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 1

161. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 1

162. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 3 | 0

163. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

164. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

165. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

166. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

167. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 1

168. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

169. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

170. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at week 24
Time Frame: Follow-up phase - Week 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

171. Secondary Outcome: Participants With Grade 1 AST Level
Description: Participants with grade 1 (1.25 - 2.5 x ULN) aspartate transaminase (AST) level at week 28
Time Frame: Follow-up phase - Week 28
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0

172. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

173. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

174. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

175. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

176. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

177. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

178. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

179. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 1 | 0

180. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

181. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

182. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

183. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

184. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

185. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

186. Secondary Outcome: Participants With Grade 2 ALT Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) alanine transaminase (ALT) level at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

187. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

188. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

189. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

190. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

191. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

192. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

193. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

194. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

195. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

196. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

197. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

198. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 1 | 0

199. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 2 | 0

200. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at week 24
Time Frame: Follow-up phase - Week 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

201. Secondary Outcome: Participants With Grade 2 AST Level
Description: Participants with grade 2 (2.6 - 5.0 x ULN) aspartate transaminase (AST) level at week 28
Time Frame: Follow-up phase - Week 28
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

202. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

203. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

204. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

205. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

206. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

207. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

208. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

209. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

210. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

211. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

212. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

213. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

214. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

215. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

216. Secondary Outcome: Participants With Grade 3 ALT Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) alanine transaminase (ALT) level at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

217. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

218. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

219. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

220. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

221. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

222. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

223. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

224. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

225. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

226. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

227. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

228. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

229. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

230. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at week 24
Time Frame: Follow-up phase - Week 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

231. Secondary Outcome: Participants With Grade 3 AST Level
Description: Participants with grade 3 (5.1 - 10.0 x ULN) aspartate transaminase (AST) level at week 28
Time Frame: Follow-up phase - Week 28
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 1

232. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

233. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

234. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

235. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

236. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

237. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

238. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

239. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

240. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

241. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

242. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

243. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine aminotransferase (ALT) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

244. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

245. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at week 20
Time Frame: Follow-up phase - Week 20
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

246. Secondary Outcome: Participants With Grade 4 ALT Level
Description: Participants with grade 4 (> 10 x ULN) alanine transaminase (ALT) level at week 24
Time Frame: Follow-up phase - Week 24
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 1

247. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 1
Time Frame: Treatment phase - Day 1
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

248. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 2
Time Frame: Treatment phase - Day 2
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

249. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 3
Time Frame: Treatment phase - Day 3
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

250. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 4
Time Frame: Treatment phase - Day 4
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

251. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 5
Time Frame: Treatment phase - Day 5
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

252. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 8
Time Frame: Treatment phase - Day 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

253. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 11
Time Frame: Treatment phase - Day 11
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

254. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 16
Time Frame: Treatment phase - Day 16
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

255. Secondary Outcome: Participants With Grade 4 AST Level
Description: Proportion of grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 24
Time Frame: Treatment phase - Day 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

256. Secondary Outcome: Participants With Grade 4 AST Level
Description: Proportion of grade 4 (> 10 x ULN) aspartate transaminase (AST) level at day 28
Time Frame: Treatment phase - Day 28
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

257. Secondary Outcome: Participants With Grade 4 AST Level
Description: Proportion of grade 4 (> 10 x ULN) aspartate transaminase (AST) level at week 8
Time Frame: Follow-up phase - Week 8
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

258. Secondary Outcome: Participants With Grade 4 AST Level
Description: Proportion of grade 4 (> 10 x ULN) aspartate transaminase (AST) level at week 12
Time Frame: Follow-up phase - Week 12
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

259. Secondary Outcome: Participants With Grade 4 AST Level
Description: Proportion of grade 4 (> 10 x ULN) aspartate transaminase (AST) level at week 16
Time Frame: Follow-up phase - Week 16
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

260. Secondary Outcome: Participants With Grade 4 AST Level
Description: Proportion of grade 4 (> 10 x ULN) aspartate transaminase (AST) level at week 24
Time Frame: Follow-up phase - Week 24
Population: Participants who received intervention
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 20 | 18
Participants | 0 | 0

261. Secondary Outcome: Participants With Grade 4 AST Level
Description: Participants with grade 4 (> 10 x ULN) aspartate transaminase (AST) level at week 28
Time Frame: Follow-up phase - Week 28
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
Number analyzed (Participants) | 19 | 18
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | GS-5734 100mg Given Intravenously Daily for 5 Days | Normal Saline Given Intravenously Daily for 5 Days
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/18
Other Adverse Events (participants affected / at risk) | 15/20 | 15/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GS-5734 100mg Given Intravenously Daily for 5 Days (N=20) | Normal Saline Given Intravenously Daily for 5 Days (N=18)
Dizziness (Cardiac disorders) | 1 | 2
Eye pain (Eye disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 2 | 1
Fatigue (General disorders) | 0 | 1
Infusion site pain (General disorders) | 3 | 5
Decreased appetite (Metabolism and nutrition disorders) | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 7
Tremor (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/82/NCT02818582/Prot_SAP_000.pdf